CLINICAL TRIAL: NCT04638764
Title: Resistance Training in Coronary Artery Disease and Heart Failure Patients Undergoing Cardiac Rehabilitation
Brief Title: Resistance Training in Cardiovascular Disease Patients
Acronym: RT in CVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital Murska Sobota (Other)
Collaborators: University of Ljubljana (Other); University of Primorska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GH-MS-CVD-RT
Record Dates: First submitted 2020-10-29; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease; Heart Failure With Reduced Ejection Fraction
Keywords: resistance training; coronary artery disease; heart failure; hemodynamic response; cardiac rehabilitation; aerobic training
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Intervention Model Description: Cluster randomisation with three parallel intervention groups
Masking Description: Baseline and post-training measurement will be performed by experienced research nurse and physiotherapist, which will not participate in intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic interval training with high loads resistance training (Active Comparator): Patient to be randomised into "combined aerobic training with high loads resistance training group".
  Interventions: Other: Aerobic interval training combined with high intensity resistance training
- Aerobic interval training with low loads resistance training (Active Comparator): Patient to be randomised into "combined aerobic training with low loads resistance training group".
  Interventions: Other: Aerobic interval training combined with low intensity resistance training
- Aerobic interval training (Active Comparator): Patient to be randomised into "aerobic training training group".
  Interventions: Other: Aerobic interval training

INTERVENTIONS:
Other: Aerobic interval training combined with high intensity resistance training — Patients enrolled in arm of the study will perform 12 weeks of combined aerobic interval training (5 intervals of cycling at the intensity of 50 %-80% of peak power obtained at baseline cardiopulmonary testing) combined with high intensity resistance training (3 sets of leg press at the intensity of 70 %- 80 % of one repetition maximum (1-RM)).
  Other Names: Aerobic and high intensity strength training
  Arms: Aerobic interval training with high loads resistance training
Other: Aerobic interval training combined with low intensity resistance training — Patients enrolled in arm of the study will perform 12 weeks of combined aerobic interval training (5 intervals of cycling at the intensity of 50 %-80% of peak power obtained at baseline cardiopulmonary testing) combined with high intensity resistance training (3 sets of leg press at the intensity of 30 %- 40 % 1-RM).
  Other Names: Aerobic and low intensity strength training
  Arms: Aerobic interval training with low loads resistance training
Other: Aerobic interval training — Patients enrolled in arm of the study will perform 12 weeks of aerobic interval training (5 intervals of cycling at the intensity of 50 %-80% of peak power obtained at baseline cardiopulmonary testing).
  Other Names: Aerobic training
  Arms: Aerobic interval training

SUMMARY:
In this study coronary artery disease patients and patients with heart failure will be randomly assigned to three training groups: combined aerobic interval training with high intensity resistance training, combined aerobic interval training with low intensity resistance training and aerobic interval training.

DETAILED DESCRIPTION:
Exercise-based cardiac rehabilitation programmes have predominantly used aerobic-dynamic exercise modalities, whereas resistance training have been discouraged in patients with cardiovascular disease, due to safety concerns related to cardiovascular response (heart rate and blood pressure) during the exertion. Contrary to such concerns, recent hemodynamic studies have reported lower blood pressure and heart rate during higher intensity resistance training (>70 % 1-RM) compared to lower intensity resistance training (>40 % 1-RM). Furthermore, the latest meta analysis have demonstrated that combined resistance training with standard aerobic interval training has been superior than aerobic training alone in several aspects of health.

However, there is still huge heterogeneity in training intervention design, also there still lacks studies to further elucidate the effects of high intensity resistance training combined with aerobic training on physical performance (aerobic capacity, muscle strength, balance), body composition, quality of life, morbidity, mortality, etc. Therefore, the aim of this study was to examine the effects of high (70%-80 % 1-RM) versus low loads (30%- 40 % 1-RM) resistance training in combination with aerobic interval cycling (50 % -80% of baseline peak Power output) in coronary artery disease patients and patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with documented CAD with clinical event (>1 month after acute coronary syndrome and/or percutaneous coronary intervention) or coronarography and/or
* Stable Heart Failure patients with documented reduced ejection fraction (>40-45 %)
* age >18 years
* NYHA class I-III
* Cardiopulmonary exercise test without ECG abnormalities

Exclusion Criteria:

* Unstable CHD
* Decompensated HF
* Uncontrolled arrhythmias
* Severe and symptomatic aortic stenosis
* Acute myocarditis, endocarditis, or pericarditis
* Aortic dissection
* Marfan syndrome
* Musculoskeletal limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-11-23 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-11-26 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal aerobic capacity | Change in maximal aerobic capacity at 12 weeks compared to baseline
  Measured as change in VO2 max (ml/kg/min)
Change in Maximal voluntary contraction of knee extensors | Change in maximal isometric torque at 12 weeks compared to baseline
  Measured as change in maximal isometric torque of knee extensors

SECONDARY OUTCOMES:
Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Change in HOMA-IR at 12 weeks compared to baseline
  Measured as change in HOMA IR (%)
Change in glucose levels | Change in glucose levels at 12 weeks compared to baseline
  Measured as change in glucose levels (mmol/L)
Change in insulin levels | Change in insulin levels at 12 weeks compared to baseline
  Measured as change in insulin levels
Change in systolic blood pressure during high and low load resistance exercise | Change of systolic blood pressure during resistance exercise compared to baseline (pre-exercise) within the first and the last week of the intervention
  Measured as change in systolic blood pressure during resistance exercise compared to baseline (pre-exercise) values
Change in diastolic blood pressure during high and low load resistance exercise | Change of diastolic blood pressure during resistance exercise compared to baseline (pre-exercise) within the first and the last week of the intervention
  Measured as change in diastolic blood pressure during resistance exercise compared to baseline (pre-exercise)
Change in heart rate during high and low load resistance exercise | Change of heart rate during resistance exercise compared to baseline (pre-exercise) within the first and the last week of the intervention
  Measured as change in heart rate during resistance exercise compared to baseline (pre-exercise)
Change in rating of perceived exertion during high and low load resistance exercise | Change of rating of perceived exertion (score 0-10, 0-no exertion, 10-maximal exertion) during resistance exercise compared to baseline (pre-exercise) within the first and the last week of the intervention
  Measured as change of rating of perceived exertion (0-10) during resistance exercise compared to baseline (pre-exercise)
Change in Short Physical Performance Battery (SPPB) total score | Change in the Short Physical Performance battery test total score (0-the worse outcome, 12- the best outcome) after 12 weeks compared to baseline
  Measured as change in points of the SPPB after 12 weeks compared to baseline
Change in time of the "Up and Go" test | Change in seconds of the "Up and Go" test after 12 weeks compared to baseline
  Measured as change of time (s) in "Up and Go" test
Change in Grip strength test (kg) | Change in kg of Grip strength test after 12 weeks compared to baseline
  Measured as change of kg in Grip strength test
Change in Arm curl test (number of repetitions) | Change in number of repetitions of the Arm curl test after 12 weeks compared to baseline
  Measured as change of number of repetitions in Arm curl test
Change in time of the Sit to stand test | Change in seconds of the Sit to stand test after 12 weeks compared to baseline
  Measured as change in time (s) of the Sit and stand test
Change in One Leg Heel Raise test (number of repetitions) | Change in number of repetitions of One leg heel raise test after 12 weeks compared to baseline
  Measured as change of number of repetitions in One leg heel raise test
Change in total energy expenditure | Change in kcal after 12 weeks compared to baseline
  Measured as change in kcal using accelerometry data
Change in sedentary activity level | Change in minutes of sedentary activity after 12 weeks compared to baseline
  Measured as change in minutes spent in sedentary activity level using accelerometry data
Change in moderate to vigorous physical activity level | Change in minutes of moderate to vigorous physical activity after 12 weeks compared to baseline
  Measured as change in minutes spent in moderate to vigorous physical activity level using accelerometry data
Change in the Back Scratch test | Change in cm of the Back Scratch test after 12 weeks compared to baseline
  Measured as change in cm of the Back Scratch test
Change in the Chair Sit and Reach test | Change in cm of the Chair sit and Reach test after 12 weeks compared to baseline
  Measured as change in cm of the Chair Sit and Reach test
Change in Stork balance test | Change in seconds of the Stork balance test after 12 weeks compared to baseline
  Measured as change in seconds of the Stork balance test
Change in Short form Health related quality of life questionnaire (SF-12) | Change in score of the Short form 12 items health related questionnaire (12 points -the lowest score, 47 points the highest score) after 12 weeks compared to baseline
  Measured as change in score of the SF-12
Change in Patients health questionnaire score (PHQ-9) | Change in score of the Patients health 9-item questionnaire (0 points-the best outcome, 27 points-the worse outcome) after 12 weeks compared to baseline
  Measured as change in points of PHQ-9 questionnaire
Change in Respiratory Exchange Ratio (RER) | Change in % after 12 weeks compared to baseline
  Measured as percent change of RER during cardiopulmonary exercise test
Change in Ve/VCO2 slope ratio | Change in ratio of VE/VCO2 slope after 12 weeks compared to baseline
  Measured as change in VE/VCO2 slope
Change in Tumor necrosis factor alpha (TNF-alpha) level | Change in TNF-alpha level after 12 weeks compared to baseline
  Measured as change in TNF-alpha
Change in Interleukin 6 (IL-6) level | Change in IL-6 level after 12 weeks compared to baseline
  Measured as change in IL-6 level
Change in Human Growth hormone (hGH) level | Change in hGH level after 12 weeks compared to baseline
  Measured as change in hGH level
Change in Insulin like Growth Factor 1 (IGF-1) | Change in IGF-1 level after 12 weeks compared to baseline
  Measured as change in IGF-1 level
Change in N-terminal-pro brain natriuretic peptide (NT-proBNP) | Change in NT-proBNP level after 12 weeks compared to baseline
  Measured as change in NT-proBNP level

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainščak, MD, PhD, Principal Investigator — General Hospital Murska Sobota; University of Ljubljana, Faculty of Medicine; Tim Kambič, MKin, Principal Investigator — General Hospital Murska Sobota; University of Ljubljana, Faculty of Sport
Locations (1):
- Division of Cardiology, General Hospital Murska Sobota, Murska Sobota, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kambic T, Bozic Mijovski M, Jug B, Hadzic V, Lainscak M. Insulin resistance, lipids and body composition in patients with coronary artery disease after combined aerobic training and resistance training: a randomised, controlled trial. Diabetol Metab Syndr. 2023 Mar 15;15(1):47. doi: 10.1186/s13098-023-01017-w. PMID 36918949
- [Derived] Kambic T, Sarabon N, Hadzic V, Lainscak M. Physical activity and sedentary behaviour following combined aerobic and resistance training in coronary artery disease patients: A randomised controlled trial. Int J Cardiol. 2023 Jan 1;370:75-79. doi: 10.1016/j.ijcard.2022.10.157. Epub 2022 Oct 29. PMID 36367488
- [Derived] Kambic T, Sarabon N, Lainscak M, Hadzic V. Combined resistance training with aerobic training improves physical performance in patients with coronary artery disease: A secondary analysis of a randomized controlled clinical trial. Front Cardiovasc Med. 2022 Aug 24;9:909385. doi: 10.3389/fcvm.2022.909385. eCollection 2022. PMID 36093154
- [Derived] Kambic T, Sarabon N, Hadzic V, Lainscak M. Effects of high-load and low-load resistance training in patients with coronary artery disease: rationale and design of a randomised controlled clinical trial. BMJ Open. 2021 Jul 22;11(7):e051325. doi: 10.1136/bmjopen-2021-051325. PMID 34301669
- [Derived] Kambic T, Hadzic V, Lainscak M. Hemodynamic Response to High- and Low-Load Resistance Exercise in Patients with Coronary Artery Disease: A Randomized, Crossover Clinical Trial. Int J Environ Res Public Health. 2021 Apr 8;18(8):3905. doi: 10.3390/ijerph18083905. PMID 33917770